CLINICAL TRIAL: NCT01451346
Title: B.Infantis 35624 in Patients With Mild to Moderate Chronic Plaque Psoriasis -a Pilot Study
Brief Title: Study in Patients With Mild to Moderate Psoriasis
Acronym: AH-PSR-01
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alimentary Health Ltd (Industry)
Collaborators: Whately-Smith Ltd, King's Langley,UK (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Psoriasis Pilot Study; AH-PSR-01 (Registry Identifier: Clinicaltrials.gov)
Record Dates: First submitted 2011-10-03; First posted 2011-10-13 (Estimated); Last update posted 2011-10-13 (Estimated); Status verified 2011-10

CONDITIONS: Psoriasis
Keywords: Pilot study
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo sachets contained 5 grams of Maltodextrin only.
  Interventions: Dietary Supplement: B. Infantis 35624
- B Infantis 35624 (Experimental): Each 5gram freeze-dried powder contained ≥1*1010 Colony forming units (CFU) of B. infantis 35624/sachet.
  Interventions: Dietary Supplement: B. Infantis 35624

INTERVENTIONS:
Dietary Supplement: B. Infantis 35624 — One sachet daily for 12 weeks

SUMMARY:
This was a randomized, double blind,fixed dose, placebo controlled, parallel-group pilot study to obtain data on size and variance of treatment effects in subjects with mild to moderate Psoriasis.

DETAILED DESCRIPTION:
This was a randomized, double blind,fixed dose, placebo controlled, parallel-group pilot study to obtain data on size and variance of treatment effects in subjects with mild to moderate Psoriasis. The target sample size of 60 was selected as a practical figure for recruitment purposes in one centre over 3 months.After a 2 week washout during which only emollients were applied to their psoriasis, patients attended for baseline assessment of psoriasis severity and blood tests.Subjects attended every 4 weeks for 12 weeks for clinical assessment and blood tests.Each patient once eligible{see inclusion & exclusion criteria} was allocated to either active treatment or placebo in identical packing for a total of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with mild to moderate psoriasis as defined by the clinician,
* Has a Psoriasis Area and Severity Index{PASI} of less than 20,
* Male or female subjects,
* Aged between 18-60 years of age,
* Non-pregnant female and must agree to use adequate method of contraception during the study,
* Is capable of giving written informed consent prior to study entry,
* Be willing to refrain from taking dietary supplements or other foods that contain fermented live bacteria within 1 month prior to treatment and during the study,
* Have not participated in a clinical drug study or used an investigational new drug during the past previous 30 days,
* Clinical Chemistry and haematology results from Visit 1 are within normal limits,
* Be willing to refrain from using any topical psoriactic cream 2 weeks prior to treatment and during the study.

Exclusion Criteria:

* Are less than 18 years of age, and not more than 60 years of age,
* History of sensitivity to lactose [eg, lactose intolerance] or other dairy products,
* History of consumption of probiotics,1 month prior to treatment,
* Being treated with steroids 2 weeks prior to entry, Diseases of the gastrointestinal tract,liver,pancreas and biliary tree[eg;gastritis,symptomatic gall stones,duodenal ulcer,gastroenteritis,diverticulitis.] Exceptions include haemorrhoids,hiatus hernia and asymptomatic gall stones.
* History of major gastric,hepatic,pancreatic or intestinal surgery or perforation,excluding cholescystectomy,appendicectomy,haemorrhoidectomy or polypectomy.
* Recent unexplained rectal bleeding and/or significant unexplained weight loss.
* Antibiotic use within one month prior to Visit 1. have a significant acute or chronic coexisting illness{cardiovascular,gastrointestinal,immunological}or a condition, which contraindicates,in the investigators judgement entry to the study.
* Patients with Diabetes Mellitus.
* Individuals who, in the opinion of the investigator, are considered to be poor clinical attendees or unlikely for any reason to be able to comply with the trial.
* Subjects currently receiving treatment involving experimental drugs.
* If a subjects has been in a recent experimental trial,must be not less than 30 days prior to this study.
* Have a concomitant end stage organ disease eg; cardiovascular,hepatic,pulmonary,renal,which , in the Investigators judgement,contraindicates participation in the study.
* Have a history of malignancy in the past 5 years with the exception of Basal Cell Carcinoma.
* Evidence of alcohol or drug abuse.
* Evidence of unstable forms of psoriasis,including guttate, erthrodermic , exfoliative or pustular psoriasis.
* Evidence of other inflammatory skin disease that may confound the evaluation of psoriasis.
* Has had systematic antipsoriatic treatment or PUVA therapy within the previous 4 weeks.
* Subject who has had UVB therapy with the previous 2 weeks.
* If the subjects scores >20% on the PASI.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2008-01; Primary Completion 2008-04 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Change in the Psoriasis area and severity index between baseline and end of feeding | At 12 weeks
  The PASI score stands for Psoriasis Area and Severity Index. This tool allows researchers to put an objective number on what would otherwise be a very subjective idea: how bad is a person's psoriasis. To make up the score, the three features of a psoriatic plaque (redness) scaling and thickness are each assigned a number from 0 to 4 with 4 being worst. Then the extent of involvement of each region of the body is scored from 0 to 6. Adding up the scores give a range of 0 to 72

SECONDARY OUTCOMES:
Psoriasis Disability Index[PDI} | at 12 weeks
  The Psoriasis Disability Index questionnaire is designed for use in adults, i.e. patients over the age of 16. It is self explanatory and can be handed to the patient who is asked to fill it in without the need for a detailed explanation. It is usually completed in three or four minutes.
  There are two possible alternative formats of the PDI. One uses visual analogue scales for each answer, the other uses tick box choices for each answer

CONTACTS AND LOCATIONS:
Overall Officials: Liam O Mahony, Dr., Study Director — Alimentary Health Ltd
Locations (1):
- Alimentary Health Ltd, Cork, Ireland